CLINICAL TRIAL: NCT02005302
Title: Study of Vitamin D2 Virus 1,25(OH)2-Vitamin D3 and Normal Protein Diet Virus Low Protein Diet in the Treatment of CKD-MBD and Malnutrition for Progressive CKD Patients
Brief Title: Optimizing Treatment Programs for Chronic Kidney Disease-mineral and Bone Disorder and Malnutrition
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wenhu Liu (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, Wenhu Liu, Professor, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJFH-EC/2013-076; D131100004713001 (Other Grant/Funding Number: Beijing Municipal Science and Technology Commission)
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Vitamin D Deficiency; Malnutrition
Keywords: chronic kidney disease; mineral and bone disease; Malnutrition; Vitamin D; low protein diet
MeSH Terms: conditions — Vitamin D Deficiency; Malnutrition; Renal Insufficiency, Chronic; Calcinosis; Bone Diseases | interventions — Ergocalciferols; Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D2 Treatment (Experimental)
  Interventions: Drug: Vitamin D2
- 1,25(OH)2 Vitamin D3 (Active Comparator)
  Interventions: Drug: 1,25(OH)2 Vitamin D3
- low protein diet (Experimental)
  Interventions: Dietary Supplement: low protein diet
- normal protein diet (Active Comparator)
  Interventions: Dietary Supplement: normal protein diet

INTERVENTIONS:
Drug: 1,25(OH)2 Vitamin D3 — Oral 1,25(OH)2 Vitamin D3 by 0.25 microgram once daily at start and regulate the dose according to the changes of blood levels of 25(OH)Vit D, calcium, phosphorus, and intact parathyroid hormone.
  Other Names: Active Vit D3
  Arms: 1,25(OH)2 Vitamin D3
Drug: Vitamin D2 — Oral Vit D2 1.25mg(50,000 unit) once weekly as a start and maintain 1.25mg(50,000 unit) once monthly according to the blood 25(OH)vitamin D level.
  Other Names: Vit D2
  Arms: Vitamin D2 Treatment
Dietary Supplement: low protein diet — Using nutritious software to make meals recipes and give dietary guidance for patients to reach the DPI goal of 0.6g-0.8g/kg/d.
  Arms: low protein diet
Dietary Supplement: normal protein diet — Using nutritious software to make meals recipes and give dietary guidance for patients to reach the DPI goal of more than 0.8g/kg/d.
  Arms: normal protein diet

SUMMARY:
Multi-center, prospective, randomized, controlled study to verify the clinical effectiveness of K / DOQI guidelines. The efficiency and safety of Vitamin D2 and low protein diet treatment for prevention and treatment of CKD-MBD and malnutrition in CKD3-5 (ND) patients.

DETAILED DESCRIPTION:
This study will enroll chronic kidney disease patients, stage 3 to 5ND, who have chronic kidney disease mineral and bone disease (CKD-MBD) and malnutrition as defined by Kidney Disease Improvement Global Outcome (KDIGO) Guidelines. Patients in five centers will be randomized. A total of 600 patients will be enrolled, 150 patients receiving Vitamin D2 treatment virus 150 patients receiving calcitriol treatment, and another 150 patients receiving low protein diet virus 150 patients receiving normal protein diet. Outcomes will be assessed as proportion of patients achieving target blood levels on calcium, phosphorus, parathyroid hormone, 25 hydroxyvitamin D, albumin and hemoglobin. Other outcomes will also be assessed, which include secondary hyperparathyroidism (sHPT), vascular calcification, cardiovascular diseases, nutritional status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18-80 years.
* Patients with chronic kidney disease stage 3 to 5, and concurrent chronic kidney disease mineral and bone disorder and malnutrition

Exclusion Criteria:

* Renal artery stenosis, inherent renal malformation, solitary kidney, or malignancy in urinary system.
* Active system immunity diseases.
* History of liver failure
* History of intestinal malabsorption or chronic diarrhea
* Treatment with phenobarbital, phenytoin, rifampicin, sucralfate, steroids, digoxin, or other medications that could affect vitamin D metabolism
* Primary hyperparathyroidism
* Treatment with cinacalcet or other calcimimetic within the past 6 months
* Anticipated dialysis within 6 months after randomization
* Have an unstable medical condition, defined as having been hospitalized within 30 days before screening, the expectation of recurrent hospital admissions or life expectancy of less than 6 months in the judgment of the investigator
* Subject is currently enrolled in, or fewer than 30 days have passed since subject has completed another investigational device or drug study(s); or subject is receiving another investigational agent(s).
* Current treatment with vitamin D 50,000 IU
* Using glucocorticoid or immunosuppressive agents.
* Acute renal dysfunction.
* The expected live time is less than 2 years.
* Pregnant or lactating woman.
* Suffered from acute myocardial infraction, acute congestive heart failure, or stroke in last 6 months.
* Patients whose concurrent illnesses, disability, or geographical residence would hamper attendance at required study visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The changes on the blood levels of calcium, phosphorus, and intact parathyroid (iPTH) hormone during 36 months | 36 months
  The blood levels of calcium, phosphorus,and intact parathyroid (iPTH) will be detected every three months. The values during follow-up will be compared to the baseline.
The changes on the clinical indicators of nutritional status | 36 months
  The blood levels of albumin, prealbumin, transferrin and hemoglobin will be detected every three months. The values during follow-up will be compared to the baseline.

SECONDARY OUTCOMES:
The changes of the blood 25(OH)Vitamin D level | 36 months
The changes of the quality of life | 36 months
  Assess the quality of life for patients in accordance with KDQOL-SF scale every 6 month. The values during follow-up will be compared to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhu Liu, Doctor, Principal Investigator — Nephrology Department of Beijing Friendship Hospita
Locations (5):
- China (5):
  - Beijing XuanWu Hospital, Beijing, Beijing Municipality
  - People's Liberation Army Air Force General Hospital, Beijing, Beijing Municipality
  - People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Sino-Japanese Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Friedship Hospital, Beijing, Beijing Municipality